CLINICAL TRIAL: NCT03852563
Title: Evaluation of the Safety and Efficacy of the Product Bepantol® Cream After the Dermatological Procedure in the Face.
Brief Title: A Study to Gain Information How Well Dexpanthenol Derma Cream Helps the Face Skin to Recover After Cosmetic Lasering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20577
Record Dates: First submitted 2019-02-15; First posted 2019-02-25 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Erythema; Skin Recovery
Keywords: Skin cream; Ablative lasering; Skin hydration; Consumer satisfaction; Sensorial perception
MeSH Terms: conditions — Erythema; Consumer Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women_Hemiface BAY207543 (Experimental): Adult women receive BAY207543 randomized to one hemiface and semisolid vaseline to the other hemiface after ablative skin lasering. The hemiface with BAY207543 is investigated.
  Interventions: Drug: BAY207543 (Bepanthol); Other: Semisolid vaseline
- Women_Hemiface Vaseline (Active Comparator): Adult women receive BAY207543 randomized to one hemiface and semisolid vaseline to the other hemiface after ablative skin lasering. The hemiface with vaseline is investigated.
  Interventions: Drug: BAY207543 (Bepanthol); Other: Semisolid vaseline

INTERVENTIONS:
Drug: BAY207543 (Bepanthol) — Product is applied to one hemiface.
Other: Semisolid vaseline — Product is applied to one hemiface.

SUMMARY:
In this study, researchers want to learn more about the effect of dexpanthenol cream on skin recovery and reduction of skin rash after a dermatological procedure (ablative laser) on the face for treatment of fine wrinkles, scars and open pores in adult women.

After the dermatological procedure, participants will return within 3 weeks for 4 visits to the study center to investigate the skin conditions such as redness, irritation, softness and possible side effects. In addition, study participants will be asked about their general acceptance of dexpanthenol cream.

DETAILED DESCRIPTION:
The primary objective is to evaluate the efficacy of the test product to aid skin recovery and reduction of erythema after ablative lasering on the face.

Secondary objectives comprise clinical efficacy with respect to skin hydration, softness, vitality, appearance etc. and skin recovery, consumer judgement of product performance and acceptability, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Phototypes I or II according to the Fitzpatrick scale
* Participants willing to perform the dermatological procedure (ablative laser) on the face for treatment of fine wrinkles, scars and open pores, rosacea
* Normal eye examination

Exclusion Criteria:

* Cutaneous pathologies and/or injuries as psoriasis, sensible skin, cancer of the skin, rosacea, atopic dermatitis or other medical criteria to be considered at the moment of the evaluation;
* Hyperpigmentation and cutaneous marks in the test area that intervenes with the evaluation of possible reactions
* Active cutaneous pathologies and/or injuries (local and/or disseminated) in the evaluation area
* Aesthetic or dermatological treatment in the area of evaluation up to 04 weeks before the selection
* People with entropy, ectropion, stye, conjunctivitis, uveitis or other active eye diseases
* People with corneal ulcerations, blepharitis, meibomitis, pterygium, trichiasis, distichiasis or other eye diseases of moderate or serious intensity

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Skin barrier integrity by TEWL probe | Up to 23 days
  The transepidermal water loss (TEWL) is measured in g m2 h-1 with a Tewameter TM300.
Dermic temperature by thermographic camera (FLIR) | Up to 23 days

SECONDARY OUTCOMES:
Skin properties of the participants | Up to 23 days
  Investigators assess various skin properties of the participants with a questionnaire (each scored from 1 to 5), resulting in an overall efficacy score from 8 to 55 (a higher score represents higher efficacy).
Treatment satisfaction | Up to 23 days
  Participants assess their treatment satisfaction with a questionnaire consisting of 23 items (each item is scored from 1-5) resulting in a score range of 23 to 115 (a higher score represents better treatment satisfaction).
Product evaluation | Up to 23 days
  Participants assess their sensorial perception of different product attributes (e.g. smell, absorption) with a questionnaire consisting of 7 items (each item is scored from 1-5) resulting in a score range from 7 to 35 (a higher score represents higher product satisfaction).
Number of adverse events by dermatological evaluation | Up to 23 days
Number of adverse events by ophthalmologic valuation | Up to 23 days
Severity of adverse events by dermatological evaluation | Up to 23 days
Severity of adverse events by ophthalmologic valuation | Up to 23 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medcin Instituto da Pele, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.